CLINICAL TRIAL: NCT00801931
Title: Double Umbilical Cord Blood Transplantation for Patients With Malignant and Non-Malignant Disorders
Brief Title: Double Cord Blood Transplant for Patients With Malignant and Non-malignant Disorders
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Prakash Satwani, Associate Professor of Pediatrics at the Columbia University Med, Department of Pediatrics BMT, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAC3457; CHNY-06-533 (Other: CU)
Record Dates: First submitted 2008-05-05; First posted 2008-12-04 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Leukemia; Lymphoma; Neuroblastoma; Immunodeficiencies; Anemia
Keywords: Cord Blood Transplant; Allogeneic Stem Cell Transplant
MeSH Terms: conditions — Leukemia; Lymphoma; Neuroblastoma; Immunologic Deficiency Syndromes; Anemia | interventions — Alemtuzumab; Whole-Body Irradiation; Melphalan; Busulfan; Phenytoin; fosphenytoin; fludarabine; fludarabine phosphate; Cyclophosphamide; Antilymphocyte Serum; thymoglobulin; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- A: Full Intensity with TBI (Experimental): Patients will start their pre-conditioning regimen on Day -8. Fractionated total body irradiation (TBI) will be administered twice daily for 3 days on Days -8, -7, and -6. Patients will receive Thiotepa on Days -5 and-4, Cyclophosphamide on Days -3 and -2 and- rabbit antithymocyte globulin on Days -4, -3, -2 and -1.The double cord blood infusion will be performed on Day 0. GM-CSF hematopoietic growth factor will start on Day 0. GVHD prophylaxis will consist of tacrolimus/mycophenolate mofetil (MMF).
  Interventions: Radiation: Total Body Irradiation; Drug: Cyclophosphamide; Drug: Rabbit Antithymocyte Globulin; Drug: Thiotepa
- B: Full intensity without TBI (Experimental): Patients will start their pre-conditioning regimen on Day -9. Patients will receive busulfan twice daily on Days - 8, -7, -6, and -5 and Melphalan on Days -4, -3 and -2 and rabbit antithymocyte globulin on Days -4, -3, -2 and -1 with double cord blood infusion on Day 0. Granulocyte-macrophage colony-stimulating factor (GM-CSF) hematopoietic growth factor will start on Day 0. GVHD prophylaxis will consist of tacrolimus/MMF.
  Interventions: Drug: Melphalan; Drug: Busulfan; Drug: Rabbit Antithymocyte Globulin
- C: Moderate Intensity (Experimental): Patients will start their GVHD prophylaxis with Tacrolimus on Day -8. Patients will receive busulfan twice daily on Days -8, -7, -6, and -5; fludarabine on Days -7, -6, -5, -4, -3 and -2 and alemtuzumab on Days -5, -4, -3, -2, and -1. The double cord blood infusion will be performed on Day 0. GVHD prophylaxis will consist of tacrolimus/MMF.
  Interventions: Drug: Alemtuzumab; Drug: Busulfan; Drug: Fludarabine
- D: Reduced Intensity (Experimental): Patients will start their GVHD prophylaxis with Tacrolimus on Day -6. Patients will receive busulfan twice daily on Days -6, and-5; fludarabine on Days -6, -5, -4, -3 and -2 and rabbit antithymocyte globulin on Days -4, -3, -2, and -1. The double cord blood infusion will be performed on Day 0. GVHD prophylaxis will consist of tacrolimus/MMF.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Rabbit Antithymocyte Globulin
- E: Fanconi's Anemia (Experimental): Patients will start their pre-conditioning regimen on Day -6. Patients will receive TBI as a single fraction on Day -6. Patients will receive fludarabine and cyclophosphamide on Days - 5, -4, -3, and -2 and horse antithymocyte globulin on Days -5, -4, -3, -2 and -1. The double cord blood infusion will be performed on Day 0. GVHD prophylaxis will consist of tacrolimus/MMF.
  Interventions: Radiation: Total Body Irradiation; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Horse Antithymocyte Globulin
- F: Regimen for non-malignant diseases (Experimental): Patients will begin fosphenytoin or phenytoin prophylaxis on Day -10. Patients will receive busulfan on days -9, -8, -7 and -6, cyclophosphamide on days -5, -4, -3, and -2 and rabbit antithymocyte globulin on days -4, -3, -2 and -1. The double cord blood infusion will be performed on Day 0. GVHD prophylaxis will consist of tacrolimus/MMF.
  Interventions: Drug: Busulfan; Drug: Phenytoin; Drug: Cyclophosphamide; Drug: Rabbit Antithymocyte Globulin

INTERVENTIONS:
Drug: Alemtuzumab — Each dose of alemtuzumab is to be diluted in 5% dextrose in water (D5W) or normal saling (NS) (maximum concentration: 0.3 mg/mL) for intravenous (IV) infusion over two hours.
  Other Names: Lemtrada; Campath
  Arms: C: Moderate Intensity
Radiation: Total Body Irradiation
  Other Names: TBI
  Arms: A: Full Intensity with TBI; E: Fanconi's Anemia
Drug: Melphalan — Melphalan 45mg/m2 (1.5 mg/kg IV for children <1 year of age or <10 kg) diluted in 0.9% NS to a concentration of 0.1- 0.45mg/ml, given IV over 30 minutes.
  Other Names: Alkeran
  Arms: B: Full intensity without TBI
Drug: Busulfan — (Busulfex) will be given IV in 0.9% sodium chloride or D5W to a final solution for infusion equal to 10 times the volume of diluent to Busulfex (to a concentration >0.5 mg/mL), through a central venous access device over 2 hours.
  Other Names: Busulfex; Myleran
  Arms: B: Full intensity without TBI; C: Moderate Intensity; D: Reduced Intensity; F: Regimen for non-malignant diseases
Drug: Phenytoin — Fosphenytoin can be administered in D5W or 0.9% sodium chloride to a final concentration ranging from 1.5 to 25 mg PE/ml at a rate of 1-3 mg phenytoin sodium equivalents (PE)/kg/min up to 50-150 mg PE/minute.
  Other Names: Fosphenytoin; Dilantin
  Arms: F: Regimen for non-malignant diseases
Drug: Fludarabine — Fludarabine will be given IV in 50-100 ml of D5W or 0.9% sodium chloride, over 30 minutes.
  Other Names: Fludara
  Arms: C: Moderate Intensity; D: Reduced Intensity; E: Fanconi's Anemia
Drug: Cyclophosphamide — Cyclophosphamide should be infused over one hour. The drug can be diluted in D5W, NS, or other solutions (100-250 mL) to a maximum concentration of 20 mg/mL.
  Other Names: Cytoxan; Neosar
  Arms: A: Full Intensity with TBI; E: Fanconi's Anemia; F: Regimen for non-malignant diseases
Drug: Horse Antithymocyte Globulin — Horse Antithymocyte Globulin (ATG [horse]) will be diluted in 0.9% sodium chloride or 0.45% sodium chloride for IV infusion (through an inline filter with pore size of 0.2 micrometer) to a concentration of 1-4 mg/ml and infused through a central venous catheter over 8 hours in Regimen E.
  Other Names: Atgam; ATG[horse]
  Arms: E: Fanconi's Anemia
Drug: Rabbit Antithymocyte Globulin — Rabbit Anti-Thymocyte Globulin (rabbit ATG) will be diluted in 0.9% sodium chloride or D5W for IV infusion (through an in-line filter with pore size of 0.22 micrometer) to a concentration of 0.5 mg/ml and infused through a central venous catheter over 8 hours for all doses on Days -4, -3, -2, and -1 in Regimens A, B, D and F.
  Other Names: Thymoglobulin
  Arms: A: Full Intensity with TBI; B: Full intensity without TBI; D: Reduced Intensity; F: Regimen for non-malignant diseases
Drug: Thiotepa — Thiotepa should be diluted in NS (1-5 mg/ml) and infused over 2 hrs on Days -8, -4. IV fluids should be at maintenance rate (1500 ml/m2).
  Other Names: Tepadina
  Arms: A: Full Intensity with TBI

SUMMARY:
The purpose of this study is to determine the safety and toxicity and feasibility of double umbilical cord blood transplantation (DUCBT) in patients with selected malignant and non-malignant, and to quantify the percentage and donor sources of mixed donor chimerism following DUCBT in patients with selected malignant and non-malignant disorders.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation from an human leukocyte antigen (HLA) matched related family donor is the treatment of choice for a wide variety of malignant and non-malignant disorders. Unfortunately, only 25% of potential recipients have an HLA matched related family donor, leaving approximately 75% of potential recipients requiring alternative sources of HLA matched allogeneic stem cells. One potential source of HLA matched allogeneic stem cells is from unrelated adult donors that have been identified in the national and international donor registries. However, several limitations restrict the uniform utilization of unrelated allogeneic adult donors including ethnic background of the recipient, acuity and timing of planned allogeneic transplant, availability of donor, and high risk of severe acute graft-versus-host disease (GVHD) (III/IV), among others. The investigators have recently identified a new alternative source of allogeneic stem cells, unrelated cryopreserved placental/cord blood stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for double cord blood stem cell transplant (TNC ≥ 4x107/kg of two combined units) if available single cord blood has TNC ≤4.0 x 107/kg and they lack a matched (5-6/6) family donor, a 10/10 unrelated adult donor, and/or if their disease status required emergent stem cell transplant and they could not wait 2-3 months for searching for a matched unrelated adult donor.
* Adequate renal function defined as:Serum creatinine <1.5 x normal, or Creatinine clearance or radioisotope glomerular filtration rate (GFR) >60 ml/min/m2 or >60 ml/min/1.73 m2 or an equivalent GFR as determined by the institutional normal range.
* Adequate liver function defined as:Total bilirubin <1.5 x normal, or serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase (AST)) or serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase (ALT)) <3.0 x normal
* Adequate cardiac function defined as:Shortening fraction >27% by echocardiogram, or Ejection fraction >47% by radionucleotide angiogram or echocardiogram.
* Adequate pulmonary function defined as:Uncorrected diffusing capacity of the lungs for carbon monoxide (DLCO) 50% by pulmonary function test.For children who are uncooperative, no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry >94% on room air.

Eligibility for Moderate Intensity, Reduced Intensity Regimen and Fanconi's Anemia (Regimens C, D and E)

* Adequate renal function defined as: Serum creatinine <2.0 x normal, or Creatinine clearance or radioisotope GFR 40 ml/min/m2 or >40 ml/min/1.73 m2 or an equivalent GFR as determined by the institutional normal range.
* Adequate liver function defined as:Total bilirubin <2.5 x normal, or SGOT (AST) or SGPT (ALT) <5.0 x normal
* Adequate cardiac function defined as:Shortening fraction of >25% by echocardiogram, or Ejection fraction >40% by radionucleotide angiogram or echocardiogram.
* Adequate pulmonary function defined as:Uncorrected DLCO >35% by pulmonary function test. For children who are uncooperative, no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry >94% on room air.

Exclusion Criteria:

* Females who are pregnant or breast-feeding
* Patients with documented uncontrolled infection at the time of study entry

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2007-09-06 (Actual); Primary Completion 2009-05-05 (Actual); Study Completion 2009-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Satwani, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia Presbyterian Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was only 1 subjected enrolled. The 1 subject was enrolled into Arm - Experimental: C: Moderate Intensity.
Groups:
- Experimental: C: Moderate Intensity: Patients will start their GVHD prophylaxis with Tacrolimus on Day -8. Patients will receive busulfan twice daily on Days -8, -7, -6, and -5; fludarabine on Days -7, -6, -5, -4, -3 and -2 and alemtuzumab on Days -5, -4, -3, -2, and -1. The double cord blood infusion will be performed on Day 0. GVHD prophylaxis will consist of tacrolimus/MMF.
Period: Overall Study
Arm/Group | Experimental: C: Moderate Intensity
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: There was only 1 subjected enrolled. The 1 subject was enrolled into Arm - Experimental: C: Moderate Intensity.
Arm/Group | Experimental: C: Moderate Intensity
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Graft Failure Rate
Description: Number of patients to experience graft failure.
Time Frame: Up to 2 years
Population: Not enough subjects were enrolled for data analysis.
Groups:
- All Subjects: Includes all subjects in the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

2. Primary Outcome: Response Rate (Complete and Partial Response)
Description: Response rate to each regimen will be measured.
Time Frame: Up to 2 years
Population: Not enough subjects were enrolled for data analysis.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

3. Primary Outcome: Overall Survival (OS)
Description: OS will be summarized using the Kaplan and Meier curves.
Time Frame: Up to 2 years
Population: Not enough subjects were enrolled for data analysis.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

4. Primary Outcome: Disease Free Survival (DFS)
Description: DFS will be summarized using the Kaplan and Meier curves.
Time Frame: Up to 2 years
Population: Not enough subjects were enrolled for data analysis.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Experimental: C: Moderate Intensity
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: C: Moderate Intensity (N=1)
Respiratory Failure with Cardiac Tamponade (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Led to death.

LIMITATIONS AND CAVEATS:
There was only 1 subjected enrolled. The 1 subject was enrolled into Arm - Experimental: C: Moderate Intensity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes